CLINICAL TRIAL: NCT01348984
Title: Transdermal Fentanyl Patch for Postoperative Analgesia in Total Knee Arthroplasty
Brief Title: Study of Transdermal Fentanyl Patch to Treat Postoperative Pain in Total Knee Arthroplasty
Acronym: TFP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Thepakorn Sathitkarnmanee, Faculty of Medicine, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TFP TKA
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2010-02

CONDITIONS: Postoperative Pain
Keywords: postoperative; pain score; morphine consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): group 1 = transdermal fentanyl patch
  Interventions: Drug: transdermal fentanyl patch
- group 2 (Placebo Comparator): placebo patch
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: transdermal fentanyl patch — TFP = transdermal fentanyl patch (50 microgram/hour)
  Other Names: Duragesic
  Arms: group 1
Drug: placebo patch — group 2 = placebo patch
  Other Names: Duragesic
  Arms: group 2

SUMMARY:
The purpose of this study is to determine whether transdermal fentanyl patch

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) has severe postoperative pain that prevents mobilization of patient. The best standard analgesia regimen is patient-control analgesia (PCA) which requires a PCA pump that is expensive.

Transdermal fentanyl patch (TFP)(50 mcg/hr) can release fentanyl into blood circulation at rate 50 mcg/hr for three days. It has slow onset of about 12-14 hours, so it's used to treat chronic pain, not popular for a cure of pain. If the investigators apply TFP at appropriate times, i.e. 12-14 hours before surgery, it may be used to treat acute postoperative pain.

If it can give good analgesia for TKA, it can replace PCA. The benefit is that it is much cheaper and more convenient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for TKA gave informed consent for inclusion

Exclusion Criteria:

* ASA class 3-4
* Known allergy to any of the drugs to be used, eg. TFPs ,MO
* History of substance or alcohol abuse, and tolerance or dependence on opioids
* Can not use PCA
* Contraindication for spinal anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
intravenous morphine consumption | 48 hours

SECONDARY OUTCOMES:
Pain score | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand